CLINICAL TRIAL: NCT03956706
Title: Phase I Study of Subventricular Zone Tumor Stem Cell Stereotactic Radiosurgery With Standard of Care Chemoradiation Therapy in Newly Diagnosed Malignant Gliomas (WHO III and WHO IV Astrocytomas)
Brief Title: Study of Stereotactic Radiosurgery to the Subventricular Zone in Malignant Gliomas
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no partipants enrolled and investigator left the institution
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-0794
Record Dates: First submitted 2019-05-14; First posted 2019-05-21 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Glioblastoma; Astrocytoma, Grade III; Astrocytoma, Grade IV; Malignant Glioma
Keywords: SRS; Stereotactic Radiosurgery; Glioblastoma; Astrocytoma; Grade III; Grade IV; Glioma; Malignant Glioma; Gamma Knife
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Glioma; Lymphoma, Follicular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Dose Escalation (18Gy) (Experimental): Receive additional dose of 18Gy to the subventricular zone
  Interventions: Radiation: Stereotactic Radiosurgery
- Dose Escalation (20Gy) (Experimental): Receive additional dose of 20Gy to the subventricular zone
  Interventions: Radiation: Stereotactic Radiosurgery
- Dose Escalation (22Gy) (Experimental): Receive additional dose of 22Gy to the subventricular zone
  Interventions: Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — Stereotactic radiosurgery dose escalation by either 18, 20, or 22 Gy to the subventricular zone in addition to standard of care
  Other Names: Gamma Knife

SUMMARY:
Several investigations suggest neural stem cells located in the subventricular region play an active role in promoting or even initiating cortical malignant glioma growth. Although normal appearing on neuroimaging, surgical specimens taken from this region show it contains malignant glioma stem-like cells. Some retrospective analyses found patients who received radiation therapy to this region during standard of care treatments lived longer than patients who did not.

The investigator's study hypothesizes (1) stereotactic radiosurgery of cancer stem-like cells in these regions will be well tolerated during standard of care therapy, (2) focused stereotactic radiosurgery will be more effective in destroying cancer stem cells than conventional radiation therapy, and (3) treatment will improve malignant glioma survival.

DETAILED DESCRIPTION:
Since 2005, standard treatment for malignant gliomas includes surgery as extensive as possible to reduce tumor bulk without causing deficits, followed by temozolomide chemotherapy with radiation therapy to the surgical area plus an additional 1-2 cm margin around this cavity. Despite advances in surgical techniques and radiation delivery, 80% of tumors recur at the margins of the surgery, within the regions that were treated with radiation.

In 2014, different institutions found patients lived longer if part of the brain that looked normal received radiation therapy. This region was called the "subventricular zone" and was known to contain embryonic stem cells that formed the brain. Researchers believed this region contained cancer stem cells promoting tumor survival and growth. Some studies suggested this area might even represent another reservoir of malignant tumor cells.

During participation in this clinical trial, targeted radiation to the subventricular zone is given in addition to standard of care radiation and chemotherapy. The subventricular zone is divided into four regions and one of four regions on the same side as the tumor is treated, not the whole subventricular zone. Only patients scheduled to receive six weeks of standard therapy are eligible for participation. The additional radiation therapy is delivered over the course of one day. The study is not randomized and all patients will receive the experimental treatment. Patients complete regular evaluations over the next two years to monitor toxicity, which is the main concern of this Phase I study.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in a clinical trial
* Confirmed WHO III or WHO IV malignant glioma, based upon Northwell Health neuropathology review. Outside cases must be submitted for central neuropathology review.
* Completion of major surgical debulking procedure, defined as residual tumor volume of less than 20% original mass
* Age greater than 18 years old. Children are not included because their disease behaves in a biologically distinct manner and there are already national clinical trials specific to them
* Patients will not be excluded on the basis of advanced age (i.e., >75 years old), but there will need to be an intent to deliver standard chemoradiation therapy. Patients scheduled for accelerated radiation therapy are ineligible
* Karnofsky performance status of 50 or higher. Patients may require considerable assistance and frequent medical care.
* Willingness to sign HIPAA authorization that allows the investigators to continue to obtain clinical information even if patient leaves the study institution for care elsewhere in order to collect long term outcome and toxicity data.
* Lobar tumor location (Frontal, temportal, parietal, occipital, or thalamic)

Exclusion Criteria:

* Inability to consent to participate in a clinical trial, as determined during the standard of care practice evaluation of a malignant brain tumor patient.
* Prior malignant glioma treatment less than 12 months prior to chemoradiation therapy, other than surgery with or without Gliadel wafer placement. Patients who received radiation therapy in the treatment of a lower grade malignancy (i.e., low grade glioma now transformed to WHO Grade III or WHO grade IV) are eligible as long as they are eligible for standard chemoradiation therapy and the radiation therapy delivered in the past was more than 12 months prior to planned chemoradiation therapy.
* Any localized interstitial radiotherapy treatment
* Concurrent clinical trial participation during standard of care therapy. Clinical trial participation is permitted in the event of recurrent disease.
* Nonlobar tumor location (e.g., callosal, brainstem, or cerebellar tumors)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the principal investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the proposed regimen
* Pregnancy is an exclusion criterion. Pregnant patients will not receive the study treatment. Women of childbearing age are routinely screened prior to radiation therapy administration for pregnancy. If found to be pregnant, then patient will not be offered participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-24 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Toxicity of Therapy | 24 months
  INCIDENCE OF TREATMENT-EMERGENT ADVERSE EVENTS AS DEFINED BY CTCAE criteria as well as BY steroid requirement

SECONDARY OUTCOMES:
Progression-free survival | 24 months
  PFS measured by time to recurrence as well as pattern of recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Alexis M Demopoulos, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health Brain Tumor Center, Lake Success, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee JH, Lee JE, Kahng JY, Kim SH, Park JS, Yoon SJ, Um JY, Kim WK, Lee JK, Park J, Kim EH, Lee JH, Lee JH, Chung WS, Ju YS, Park SH, Chang JH, Kang SG, Lee JH. Human glioblastoma arises from subventricular zone cells with low-level driver mutations. Nature. 2018 Aug;560(7717):243-247. doi: 10.1038/s41586-018-0389-3. Epub 2018 Aug 1. PMID 30069053
- [Background] Piccirillo SG, Spiteri I, Sottoriva A, Touloumis A, Ber S, Price SJ, Heywood R, Francis NJ, Howarth KD, Collins VP, Venkitaraman AR, Curtis C, Marioni JC, Tavare S, Watts C. Contributions to drug resistance in glioblastoma derived from malignant cells in the sub-ependymal zone. Cancer Res. 2015 Jan 1;75(1):194-202. doi: 10.1158/0008-5472.CAN-13-3131. Epub 2014 Nov 18. PMID 25406193
- [Background] Bao S, Wu Q, McLendon RE, Hao Y, Shi Q, Hjelmeland AB, Dewhirst MW, Bigner DD, Rich JN. Glioma stem cells promote radioresistance by preferential activation of the DNA damage response. Nature. 2006 Dec 7;444(7120):756-60. doi: 10.1038/nature05236. Epub 2006 Oct 18. PMID 17051156
- [Background] Chen L, Guerrero-Cazares H, Ye X, Ford E, McNutt T, Kleinberg L, Lim M, Chaichana K, Quinones-Hinojosa A, Redmond K. Increased subventricular zone radiation dose correlates with survival in glioblastoma patients after gross total resection. Int J Radiat Oncol Biol Phys. 2013 Jul 15;86(4):616-22. doi: 10.1016/j.ijrobp.2013.02.014. Epub 2013 Mar 26. PMID 23540348
- [Background] Ogura K, Mizowaki T, Arakawa Y, Ogura M, Sakanaka K, Miyamoto S, Hiraoka M. Initial and cumulative recurrence patterns of glioblastoma after temozolomide-based chemoradiotherapy and salvage treatment: a retrospective cohort study in a single institution. Radiat Oncol. 2013 Apr 23;8:97. doi: 10.1186/1748-717X-8-97. PMID 24499582